CLINICAL TRIAL: NCT05372198
Title: A Single-center, Open-label, Cohort Study of Surufatinib With or Without Immunotherapy in Patients With Advanced Colorectal Cancer Who Have Failed Front-line Antiangiogenic TKI Therapy
Brief Title: Surufatinib With or Wothout Immunotherapy for Advanced Colorectal Cancer in Later Line
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Abdominal Oncology Department，Deputy Director, Hubei Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCKY2021030
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Surufatinib Monotherapy (Experimental): Patients who met the eligibility criteria took Surufatinib 300mg qd, every 3 weeks as a cycle
  Interventions: Drug: Chohort 1: Surufatinib
- Cohort 2: Surufatinib with immunotherapy (Experimental): Patients who met the eligibility criteria took Surufatinib with immunotherapy:
  Surufatinib:250mg qd, every 3 weeks as a cycle Immunotherapy: Refer to the instructions for the use of immunotherapy, every 3 weeks as a cycle
  Interventions: Drug: Chohort 2: Immunotherapy; Drug: Chohort 2: Surufatinib

INTERVENTIONS:
Drug: Chohort 1: Surufatinib — Surufatinib 300mg, qd, every 3 weeks as a cycle
  Arms: Cohort 1: Surufatinib Monotherapy
Drug: Chohort 2: Immunotherapy — Refer to the instructions for the use of immunotherapy, every 3 weeks as a cycle
  Arms: Cohort 2: Surufatinib with immunotherapy
Drug: Chohort 2: Surufatinib — Surufatinib 250mg, qd, every 3 weeks as a cycle
  Arms: Cohort 2: Surufatinib with immunotherapy

SUMMARY:
This is a single-center, open-label, cohort clinical study to investigate the efficacy and safety of surufatinib with or without immunotherapy in patients with advanced colorectal cancer who failed front-line anti-angiogenic TKI therapy.

Patients have to received at least a second-line standard therapy or cannot tolerate other treatments, and have previously failed anti-angiogenic TKIs therapy(including but not limited to: fruquintinib/regorafenib/anlotinib) / apatinib, and are resistant to treatment, disease progression, intolerable toxicity or no continued benefit as assessed by investigator after therapy).

Patients who met the eligibility criteria are randomized 1:2 into two cohorts (cohort 1: surufatinib, cohort 2: surufatinib plus immunotherapy) to receive treatment until disease progression, death, unacceptable toxicity, withdrawal of consent by the patient, or decision by the treating physician that discontinuation would be in the patient's best interest. The primary study endpoint was PFS(progression free survival).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent has been signed；
* Age ≥ 18 years, ≤80 years；
* Histologically confirmed advanced colorectal cancer；
* Patients have to received at least a second-line standard therapy or cannot tolerate other treatments, and have previously failed anti-angiogenic TKIs therapy(including but not limited to: fruquintinib/regorafenib/anlotinib) / apatinib, and are resistant to treatment, disease progression, intolerable toxicity or no continued benefit as assessed by investigator after therapy)；
* ECOG 0-2；
* Life expectancy ≥ 12 weeks
* Patients must have adequate organ function；
* Women of childbearing age must have a negative pregnancy test within the first day of the study, and contraceptive methods should be taken during the study until 6 months after the last administration.

Exclusion Criteria:

* Have previously received surufatinib or immunotherapy;
* Have received other systemic anti-tumor therapies within 2 weeks(eg.chemotherapy or radiotherapy, immunotherapy, targeted therapy, and traditional Chinese medicine therapy);
* Participating in other drug clinical trials within 4 weeks before recruited;
* Have received major surgery within 4 weeks;
* Patients had other malignant tumors in the past 5 years or at the same time (except for the cured skin basal cell carcinoma and cervical carcinoma in situ);
* Pleural effusion or ascites causing relevant clinical symptoms , including respiratory syndrome (dyspnea≥CTC AE grade 2)；
* Clinically significant electrolyte abnormality；
* Systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 90mmHg regardless of any antihypertensive drugs；
* Patient currently has any disease or condition that affects drug absorption, or the patient cannot take surufatinib orally；
* Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI；
* Have evidence or history of bleeding tendency within 3 months or thromboembolic events within 12 months before enrollment;
* Clinically significant cardiovascular disease;
* Active or uncontrolled serious infection (≥CTCAE grade 2 infection);
* Clinical uncontrolled active infections, including human immunodeficiency virus (HIV) infection, active hepatitis B / C (HBV DNA Positive[1×104 copies/mL or >2000 IU/ml], HCV RNA positive[>1×103 copies/mL]);
* Patients have untreated central nervous system metastasis；
* Patients have not recovered from all toxicities associated with prior anti-tumor therapy ,to acceptable baseline status, or a NCI CTCAE v5.0 Grade of 0 or 1, except for alopecia, lymphopenia, and neurotoxicity of grade ≤2 due to chemotherapeutic drugs;
* Pregnant or lactating women;
* Have received blood transfusion therapy, blood products and hematopoietic factors within 14 days;
* Proteinuria ≥ 2+ (1.0g/24hr);
* There are concomitant diseases (such as severe hypertension, diabetes, thyroid disease, active infection, etc.) that seriously endanger the safety of patients or affect the completion of the study, or any laboratory abnormalities that are not suitable for participating in the clinical trial according to the judgment of the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 36 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

SECONDARY OUTCOMES:
overall survival (OS) | 36 months
  OS is the time from enrollment to death due to any cause.
objective response rate (ORR) | 36 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.
disease control rate (DCR) | 36 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
quality of life (QoL) assessed by the QLQ-C30 | 36 months
  QoL was defined as specific questionnaires can be used to evaluate the daily living ability of patients, so as to evaluate the effect of anti-tumor drug treatment In clinical research
adverse events (AE) | 36 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No